CLINICAL TRIAL: NCT00521664
Title: Prospective Randomized Trial Comparing a Prophylactic With a Therapeutic Platelet Transfusion Strategy in Two Groups: 1)in Patients With Acute Myeloid Leukemia After Intensive Chemotherapy and 2) After Autologous Blood Stem Cell Transplantation
Brief Title: A Trial Comparing a Prophylactic With a Therapeutic Platelet Transfusion Strategy in Two Groups
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Katrin Peschel, Dresden University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEI 1224/01
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Myeloid Leukemia
Keywords: proof of safety and cost effectiveness of the new therapeutic platelet transfusion strategy
MeSH Terms: conditions — Leukemia, Myeloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Therapeutic platelet transfusion (TP) strategy versus prophylactic platelet transfusion (PP) strategy. In the TP arm platelet transfusion is only required if bleeding occurs (more than petechial)or in case of pulmonary infections with or without sepsis.
  Interventions: Biological: Therapeutic platelet transfusion
- 2 (Active Comparator): In the PP arm platelet transfusion has to be performed when platelet count is below 10.000/µL in any case and when bleeding (more than petechial) occurs.
  Interventions: Biological: Prophylactic platelet transfusion

INTERVENTIONS:
Biological: Prophylactic platelet transfusion — In the PP arm platelet transfusion has to be performed when platelet count is below 10.000/µL in any case and when bleeding (more than petechial) occurs.
  Arms: 2
Biological: Therapeutic platelet transfusion — In the TP arm platelet transfusion is only required if bleeding occurs (more than petechial)or in case of pulmonary infections with or without sepsis.
  Arms: 1

SUMMARY:
The purpose of this study is to show that a therapeutic platelet transfusion strategy (i.e. platelet transfusion only in case of bleeding) needs minimally a quarter less of transfusions compared to the standard prophylactic transfusion strategy (i.e. platelet transfusion without any sign of bleeding when the platelet count is below 10.000/µL). With the experimental transfusion strategy transfusions could be safely reduced when the study hypothesis can be proven. This is the first prospective randomized study on this topic.

ELIGIBILITY:
Inclusion Criteria:

AML project

* inclusion in studies of the DSIL or OSHO group for AML
* AML M3/M3v can be included only when in complete remission
* age 16 - 80 years
* written informed consent

Autologous project

* AMl and ALL patients in first or second remission
* low grade or high grade non hodgkin lymphoma or morbus hodgkin or multiple myeloma
* conditioning regime: TBI 8-12 Gy/Cy 120 or BEAM or BU/CY or Melphalan 140-200mg/m2 or a similarly intensive chemotherapy regime
* age 16 - 65 years

Exclusion Criteria:

AML project

* known refractoriness to platelet transfusion
* known major bleeding with thrombocytopenia when the reason for bleeding is still ongoing
* known plasmatic coagulation disorder
* patient unable to give informed consent

Autologous project

* known refractoriness to platelet transfusion
* known major bleeding with thrombocytopenia when the reason for bleeding is still ongoing
* known plasmatic coagulation disorder
* patient unable to give informed consent
* patients with pulmonal or cerebral lesions due to infection or neoplasm
* patients with al-amyloidosis

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
reduction in numbers of platelet transfusion by 25 % in the experimental arm (therapeutic transfusion strategy)compared with the standard arm (prophylactic transfusion strategy) | 2010

SECONDARY OUTCOMES:
- incidence and duration of clinically relevant bleeding - numbers of red blood cell transfusion - side effects of transfusions - duration of thrombocytopenia below 10.000/µL and below 20.000/µL - duration of hospitalisation | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Ehninger, Prof., Principal Investigator — University Hospital Carl Gustav Carus Dresden
Locations (1):
- Klinikum Nürnberg Nord; Einheit für Knochenmarktransplantation; 5. Med. Klinik, Nuremberg, Germany

REFERENCES:
- [Derived] Wandt H, Schaefer-Eckart K, Wendelin K, Pilz B, Wilhelm M, Thalheimer M, Mahlknecht U, Ho A, Schaich M, Kramer M, Kaufmann M, Leimer L, Schwerdtfeger R, Conradi R, Dolken G, Klenner A, Hanel M, Herbst R, Junghanss C, Ehninger G; Study Alliance Leukemia. Therapeutic platelet transfusion versus routine prophylactic transfusion in patients with haematological malignancies: an open-label, multicentre, randomised study. Lancet. 2012 Oct 13;380(9850):1309-16. doi: 10.1016/S0140-6736(12)60689-8. Epub 2012 Aug 8. PMID 22877506